CLINICAL TRIAL: NCT07302802
Title: Efficacy of Semaglutide s.c. Once-weekly on Weight Loss and Management in Adolescents With Monogenic Obesity in Clinical Practice
Status: Recruiting | Type: Observational
Sponsor: Prof. Dr. Martin Wabitsch (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. Martin Wabitsch, Principal Investigator, University of Ulm
Organization: University of Ulm (Other)
Other Study IDs: U1111-1307-1203
Record Dates: First submitted 2025-12-10; First posted 2025-12-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Monogenic Obesity
Keywords: semaglutide; monogenic obesity
MeSH Terms: interventions — semaglutide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 68 Weeks
Biospecimen Retention: Samples With DNA — Serum, plasma, whole blood (EDTA), fat tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (6):
- Patients with biallelic variants in the LEPR, PCSK1, POMC, and MC4R gene
  Interventions: Drug: Semaglutide (administered by PDS290 pen-injector)
- Patients with monoallelic variants in the LEPR gene
  Interventions: Drug: Semaglutide (administered by PDS290 pen-injector)
- Patients with monoallelic variants in the PCSK1 gene
  Interventions: Drug: Semaglutide (administered by PDS290 pen-injector)
- Patients with monoallelic variants in the POMC gene
  Interventions: Drug: Semaglutide (administered by PDS290 pen-injector)
- Patients with monoallelic variants in the MC4R gene
  Interventions: Drug: Semaglutide (administered by PDS290 pen-injector)
- Patients with monoallelic variants in the SH2B1 gene or with 16p11.2 deletions
  Interventions: Drug: Semaglutide (administered by PDS290 pen-injector)

INTERVENTIONS:
Drug: Semaglutide (administered by PDS290 pen-injector) — Treatment with semaglutide as prescribed in routine clinical practice according to summary of product characteristics. The use of semaglutide can be categorised into two groups during enrolment period: 1. new users, or 2. current users (e.g., those continuing semaglutide treatment prescribed in routine clinical practice).

SUMMARY:
This observational study aims to assess the effect of once-weekly s.c. semaglutide 2.4 mg as an adjunct to a calorie-reduced diet and increased physical activity on weight loss, change in hunger, body composition, depression, and quality of life after 68 weeks of treatment in adolescents diagnosed with monogenic obesity in routine clinical care.

DETAILED DESCRIPTION:
The primary objective of this prospective, non-interventional observational study is to evaluate the effect of once-weekly s.c. semaglutide 2.4 mg in routine clinical care as an adjunct to a calorie-reduced diet and increased physical activity on weight loss after 68 weeks of treatment in adolescents diagnosed with monogenic obesity.

The secondary objectives of this prospective, non-interventional observation are to evaluate treatment compliance and to assess the influence of once-weekly s.c. semaglutide 2.4 mg in clinical practice on hunger score, body mass parameters, body composition, and depression score after 68 weeks of treatment in adolescents diagnosed with monogenic obesity. In addition, we will document the known parameters of safety and tolerability to determine safety and tolerability in clinical practice.

The exploratory objective of this prospective, non-interventional observation is to assess user satisfaction by measuring change in subjective hunger score, quality of life, and perceptions and attitudes regarding treatment with semaglutide in adolescents diagnosed with monogenic obesity treated in routine clinical practice with once-weekly s.c. semaglutide 2.4 mg after 68 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment with semaglutide as prescribed in routine clinical practice according to summary of product characteristics.
2. Informed consent of the patient, their parents, or legally acceptable representative (LAR) of participant and adolescent assent, as age-appropriate.
3. Age at time of signing informed consent: ≥12 to <21 years.
4. BMI ≥95th percentile as defined on sex- and age-specific BMI growth charts (CDC.gov)
5. Body weight of >60 kg.
6. Diagnosis of monogenic obesity by a Clinical Laboratory Improvement Amendments (CLIA)/ College of American Pathologists (CAP)/International Organisation for Standardization (ISO) 1518-certified laboratory using ACMG criteria as pathogenic (P), likely pathogenic (LP) and variant of uncertain significance (VUS).

Exclusion Criteria:

1. Participation in any interventional clinical trials at the time of enrolment.
2. Females of childbearing potential who are not using adequate contraceptive methods (as required by local law or practice)
3. Hypersensitivity to the active substance or to any of the excipients listed:

   * Disodium phosphate, dihydrate
   * Propylene glycol
   * Phenol
   * Hydrochloric acid (for pH adjustment)
   * Sodium hydroxide (for pH adjustment)
   * Water for injection
4. The safety and efficacy of Wegovy have not been investigated in patients:

   * treated with other products for weight management,
   * with type 1 diabetes,
   * with severe renal impairment (see section 4.2),
   * with severe hepatic impairment (see section 4.2),
   * with congestive heart failure New York Heart Association (NYHA) class IV. Use in these patients is not recommended

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged ≥12 to <21 years diagnosed with monogenic obesity, who agreed on treatment with semaglutide, are eligible for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving ≥10% BMI reduction from baseline (week 0) to week 68. | 68 weeks
  The study evaluates the effect of once-weekly subcutaneous (s.c.) semaglutide 2.4 mg administered as an adjunct to a calorie-reduced diet and increased physical activity in adolescents diagnosed with monogenic obesity. This measure focuses on weight loss effectiveness, with the goal of assessing the impact of the treatment on BMI reduction in a real-world clinical setting after 68 weeks of treatment. The study aims to provide insight into the potential of semaglutide in managing weight in this specific patient population.

SECONDARY OUTCOMES:
Secondary Endpoints for Weight and Health Parameters | 68 weeks
  The secondary endpoints of this study focus on changes in health outcomes over 68 weeks. These include body weight and BMI, measured as percentages or in kg and kg/m², with specific thresholds (e.g., 95th percentile) for age- and sex-specific BMI. Blood pressure (systolic and diastolic) is recorded in mmHg. Cholesterol levels (total, HDL, LDL, triglycerides) are assessed in mg/dL to evaluate cardiovascular risk. HbA1c (percentage), fasting glucose (mg/dL), and insulin (pmol/L) are monitored for metabolic health. ALT (IU/L) measures liver function. Changes in fat and lean mass are evaluated by DXA (kg). Weight and BMI velocity are measured in percentage points. The proportion of participants achieving ≥5% and ≥15% BMI reduction is also reported, offering insight into the treatment's effectiveness on weight and metabolic health.

CONTACTS AND LOCATIONS:
Locations (7):
- Assistance Publique-Hôpitaux de Paris (AP-HP), Trousseau Hospital Paris, Pediatric Nutrition Department, Paris, France
- Germany (3):
  - Institute for Experimental Pediatric Endocrinology, Charité Universitätsmedizin Berlin, Berlin
  - University Hospital for Children and Adolescents, Center for Pediatric Research, Medical Faculty, University of Leipzig, Leipzig
  - Division of Paediatric Endocrinology and Diabetes, Department of Paediatrics and Adolescent Medicine, Ulm University Medical Centre, Ulm
- University Medical Center Rotterdam, Erasmus MC-Sophia Children's Hospital, Rotterdam, Netherlands
- Departments of Pediatrics & Pediatric Endocrinology, Hospital Infantil Universitario Niño Jesús, Universidad Autónoma de Madrid, Madrid, Spain
- Wellcome-MRC Institute of Metabolic Science and NIHR Cambridge Biomedical Research Centre, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Due to participant confidentiality requirements under GDPR regulations, IPD will not be shared. The study design also limits data sharing at this stage

REFERENCES:
- [Background] Welling MS, de Groot CJ, Kleinendorst L, van der Voorn B, Burgerhart JS, van der Valk ES, van Haelst MM, van den Akker ELT, van Rossum EFC. Effects of glucagon-like peptide-1 analogue treatment in genetic obesity: A case series. Clin Obes. 2021 Dec;11(6):e12481. doi: 10.1111/cob.12481. Epub 2021 Jul 21. PMID 34291582
- [Background] Iepsen EW, Have CT, Veedfald S, Madsbad S, Holst JJ, Grarup N, Pedersen O, Brandslund I, Holm JC, Hansen T, Torekov SS. GLP-1 Receptor Agonist Treatment in Morbid Obesity and Type 2 Diabetes Due to Pathogenic Homozygous Melanocortin-4 Receptor Mutation: A Case Report. Cell Rep Med. 2020 Apr 21;1(1):100006. doi: 10.1016/j.xcrm.2020.100006. eCollection 2020 Apr 21. PMID 33205056
- [Background] Wabitsch M, Farooqi S, Fluck CE, Bratina N, Mallya UG, Stewart M, Garrison J, van den Akker E, Kuhnen P. Natural History of Obesity Due to POMC, PCSK1, and LEPR Deficiency and the Impact of Setmelanotide. J Endocr Soc. 2022 Apr 15;6(6):bvac057. doi: 10.1210/jendso/bvac057. eCollection 2022 Jun 1. PMID 35528826
- [Background] Courbage S, Poitou C, Le Beyec-Le Bihan J, Karsenty A, Lemale J, Pelloux V, Lacorte JM, Carel JC, Lecomte N, Storey C, De Filippo G, Coupaye M, Oppert JM, Tounian P, Clement K, Dubern B. Implication of Heterozygous Variants in Genes of the Leptin-Melanocortin Pathway in Severe Obesity. J Clin Endocrinol Metab. 2021 Sep 27;106(10):2991-3006. doi: 10.1210/clinem/dgab404. PMID 34097736
- [Background] Nordang GBN, Busk OL, Tveten K, Hanevik HI, Fell AKM, Hjelmesaeth J, Holla OL, Hertel JK. Next-generation sequencing of the monogenic obesity genes LEP, LEPR, MC4R, PCSK1 and POMC in a Norwegian cohort of patients with morbid obesity and normal weight controls. Mol Genet Metab. 2017 May;121(1):51-56. doi: 10.1016/j.ymgme.2017.03.007. Epub 2017 Mar 29. PMID 28377240